CLINICAL TRIAL: NCT07098819
Title: The eValuation of Sources of vIBRAtioN for Vibrational Shear Wave elasTography
Acronym: VIBRANT
Status: Not yet recruiting | Type: Observational
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Other Study IDs: CCR5897
Record Dates: First submitted 2025-06-26; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Head and Neck Cancer (H&Amp;Amp;N); Lymph Nodes
Keywords: vibrational shear wave elastography; ultrasound imaging
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy volunteers
  Interventions: Device: Vibrational Shear wave elastography algorithm

INTERVENTIONS:
Device: Vibrational Shear wave elastography algorithm — An algorithm that detects the propogation of shear waves in the head and neck.

SUMMARY:
Patients suffering with Head and Neck Cancer often must wait 3 months or more to know if their treatment has been effective, which can be very stressful. The investigators are developing an imaging tool that may be useful to help clinicians understand if patients need secondary treatment, surgery to remove lymph nodes in the neck, sooner. Evidence suggests that lymph nodes containing cancer are stiffer than normal lymph nodes.

The investigator's tool, vibrational shear wave elastography, measures the stiffness of tissue using shear waves. Gentle vibrations, like those of a mobile phone, applied to the skin surface can create shear waves in the body. The investigators use ultrasound imaging and an algorithm the investigators have developed to measure shear wave speed which is related to tissue stiffness. The algorithm is applied to ultrasound images using software we have written.

To help develop the software the investigators wish to explore different ways of creating shear waves in the neck and see how well the investigators can detect shear waves as they pass through tissues such as muscle, the thyroid and other glands in the neck. The investigators will recruit healthy volunteers to participate in this study. The investigators will use external vibrational sources gently placed against the neck in different positions to understand what the best approach to achieve the best measurement of tissue stiffness is. The investigators will also ask healthy volunteers to generate vibrations themselves using their vocal cords, a process called vocal fremitus. Participants will be asked utter 'aaa' sounds at different pitches, and the investigators will image the shear wave generated by the vibrating vocal cords. The investigators will also ask volunteers how comfortable they found the external vibrations and how easy or difficult they found it to utter and hold the sounds. This study is an exploratory benchmarking study of the software that will help the investigators develop our technique further, and design and build optimal equipment before testing it in patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers

Exclusion Criteria:

* Healthy volunteers who do not consider themselves to currently have normal neck mobility and feel able to lie supine with their neck supported for up to 90 minutes.
* Volunteers who are receiving treatment for diseases of the thyroid, glands, or lymph nodes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult volunteers
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Mean shear wave speed | Day 1
  Mean shear wave speed in neck tissues (thyroid gland, submandibular gland, parotid, or superficial cervical lymph nodes, adipose tissue, muscle, and cartilage) measured using VSWE software, acquired using external sources.

IPD SHARING:
Plan to Share IPD: Undecided